CLINICAL TRIAL: NCT05593159
Title: Evaluating the Clinical Performance of a Bioactive Restorative Material in Non-Carious Cervical Lesions
Brief Title: Bioactive Restorative Material in Non-Carious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-OperativeDent-02-2023
Record Dates: First submitted 2022-10-12; First posted 2022-10-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cervical Lesion
Keywords: Non-carious cervical lesions (NCCLs); Composite restorations; Bioactive Restorative Material (Cention N); Adhesive

STUDY DESIGN:
Intervention Model Description: Split mouth design; each patient will receive three restorations, one for each arm of this study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Clinical evaluation of restorations will be conducted by two trained and calibrated examiners. All examiners and patients are going to be blinded from group assignment. Allocation concealment will be done by using sequentially numbered, sealed/opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dentin Conditioning & RM-GIC (Active Comparator): Dentin Conditioning:
  After washing and drying -but not desiccating- Dentin Conditioner 20% (GC, Japan) will be applied using a cotton pellet for 20 seconds then rinsed thoroughly and gently dried.
  RM-GIC:
  RM-GIC (Fuji II LC) will be applied in <2mm incremental layers afterward light-cured for 10 sec (1,000 mW/cm2) per increment to fill the cavity.
  Interventions: Other: Dentin Conditioning; Other: RM-GIC
- 1-step adhesive & Cention N (Experimental): 1-step adhesive: A universal adhesive system (Tetric® N-Bond Universal) will be applied on both enamel and dentin and gently scraped for 20 sec, then dispersed with oil-free gentle air stream, then light-cured for 10 sec (1,000 mW/cm2).
  Cention N:
  The cavity will be restored using cention N followed by light curing for 10sec (1,000 mW/cm2)
  Interventions: Other: 1-step adhesive; Other: Cention N
- Dentin roughness & Gingival retentive groove preparation & Cention N (Experimental): Dentin roughness:
  Using a round carbide bur size 14/16, (H1SEM.204.014 VPE5 or H1SEM.204.016 VPE 5, Komet Dental, Lemgo, Germany) on a low-speed handpiece. (No bevel preparation will be made)
  Gingival retentive groove preparation:
  Using size-010 round carbide bur (H1SEM.205.010 VPE 5, Komet Dental, Lemgo, Germany) on a low-speed handpiece.
  Cention N:
  The cavity will be restored using cention N followed by light curing for 10sec (1,000 mW/cm2)
  Interventions: Other: Cention N; Other: Dentin roughness; Other: Gingival retentive groove preparation

INTERVENTIONS:
Other: Dentin Conditioning — After washing and drying -but not desiccating- Dentin Conditioner 20% (GC, Japan) will be applied using a cotton pellet for 20 seconds then rinsed thoroughly and gently dried
  Arms: Dentin Conditioning & RM-GIC
Other: RM-GIC — RM-GIC (Fuji II LC) will be applied in <2mm incremental layers afterword light-cured for 10 sec (1,000 mW/cm2) per increment to fill the cavity.
  Arms: Dentin Conditioning & RM-GIC
Other: 1-step adhesive — A universal adhesive system (Tetric® N-Bond Universal) will be applied on both enamel and dentin and gently scraped for 20 sec, then dispersed with oil-free gentle air stream, then light-cured for 10 sec (1,000 mW/cm2).
  Arms: 1-step adhesive & Cention N
Other: Cention N — The cavity will be restored using cention N followed by light curing for 10sec (1,000 mW/cm2)
  Arms: 1-step adhesive & Cention N; Dentin roughness & Gingival retentive groove preparation & Cention N
Other: Dentin roughness — Using a round carbide bur size 14/16, (H1SEM.204.014 VPE5 or H1SEM.204.016 VPE 5, Komet Dental, Lemgo, Germany) on a low-speed handpiece. (No bevel preparation will be made)
  Arms: Dentin roughness & Gingival retentive groove preparation & Cention N
Other: Gingival retentive groove preparation — Using size-010 round carbide bur (H1SEM.205.010 VPE 5, Komet Dental, Lemgo, Germany) on a low-speed handpiece.
  Arms: Dentin roughness & Gingival retentive groove preparation & Cention N

SUMMARY:
Evaluating the clinical performance of a bioactive restorative materiel (Cention N) placed in non-carious cervical lesions (NCCLs) with no preparation and 1-step adhesive system or, with preparing a gingival retentive groove and no adhesive system.

DETAILED DESCRIPTION:
Cention N is a relatively new restorative material that is known to be the first commercially available bioactive resin composite. The manufacturing company recommends using Cention N with 1-step adhesive system in non-retentive cavities, or with no adhesive system in retentive cavity preparations.

This study was designed to evaluate the clinical performance of this material in non-carious cervical lesions by comparing it to RM-GIC (Fuji II LC).

Information about oral and tooth brushing habits along with detailed information about the characteristics of each NCCL, gingival status, and preoperative sensitivity will be collected for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* with at least 20 teeth under occlusion
* Should have three or more NCCLs which share the characteristics of being deeper than 1 mm, and involve both the enamel and dentin of vital teeth without mobility

Exclusion Criteria:

* Poor oral hygiene
* Severe periodontitis
* Severe bruxism habits
* Xerostomia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in retention rate | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by Modified United States Public Health Service criteria (USPHS) Alpha: Retained. Bravo: Partially retained. Charlie: Missing.

SECONDARY OUTCOMES:
Change in marginal adaptation | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: Restoration is continuous with existing anatomic form. Bravo: Detectable V-shaped defect in enamel only. Catches explorer going both ways. Charlie: Detectable V-shaped defect to dentin-enamel junction.
Change in restoration fracture | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: None. Bravo: Small chip, but Clinically acceptable. Charlie: Failure due to bulk restorative fracture.
Change in marginal discoloration | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: No discoloration along the margin. Bravo: Slight and superficial staining (removable, usually localized). Charlie: Deep staining cannot be polished away.
Change in anatomic form | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: Appropriate contour. Bravo: Slightly over/under contoured. Charlie: Unacceptably over/under contoured
Change in surface texture | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: Enamel-like surface. Bravo: Surface rougher than enamel (clinically acceptable). Charlie: Surface unacceptably rough.
Change in secondary caries | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: No evidence of caries contiguous with the margin. Charlie: Evidence of presence of caries.
Change in post-operative sensitivity with stimulation | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by Modified visual analog scale (VAS).
Change in post-operative sensitivity without stimulation | Baseline: 1 day, follow-ups after 1 week, 1 month, 3 months, 6 months, 9 months, 1 year
  Rated by Modified visual analog scale (VAS).
Change in patient satisfaction | Baseline: 1 week, follow-ups after 3 months, 6 months, 9 months, 1 year
  Rated by modified USPHS. Alpha: Patient is totally satisfied. Bravo: Patient has esthetic complains, or complains related to the inability to chew comfortably. Charlie: Patient is completely unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Hussam Milly, PhD, Study Director — Milly
Locations (1):
- Restorative Dentistry, Faculty of Dental Medicine, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bezerra IM, Brito ACM, de Sousa SA, Santiago BM, Cavalcanti YW, de Almeida LFD. Glass ionomer cements compared with composite resin in restoration of noncarious cervical lesions: A systematic review and meta-analysis. Heliyon. 2020 May 21;6(5):e03969. doi: 10.1016/j.heliyon.2020.e03969. eCollection 2020 May. PMID 32462087
- [Result] Francois P, Fouquet V, Attal JP, Dursun E. Commercially Available Fluoride-Releasing Restorative Materials: A Review and a Proposal for Classification. Materials (Basel). 2020 May 18;13(10):2313. doi: 10.3390/ma13102313. PMID 32443424
- [Result] Francois P, Remadi A, Le Goff S, Abdel-Gawad S, Attal JP, Dursun E. Flexural properties and dentin adhesion in recently developed self-adhesive bulk-fill materials. J Oral Sci. 2021 Mar 31;63(2):139-144. doi: 10.2334/josnusd.20-0448. Epub 2021 Feb 17. PMID 33597335
- [Result] Kim SY, Lee KW, Seong SR, Lee MA, Lee IB, Son HH, Kim HY, Oh MH, Cho BH. Two-year clinical effectiveness of adhesives and retention form on resin composite restorations of non-carious cervical lesions. Oper Dent. 2009 Sep-Oct;34(5):507-15. doi: 10.2341/08-006C. PMID 19830963
- [Result] Loguercio AD, Luque-Martinez IV, Fuentes S, Reis A, Munoz MA. Effect of dentin roughness on the adhesive performance in non-carious cervical lesions: A double-blind randomized clinical trial. J Dent. 2018 Feb;69:60-69. doi: 10.1016/j.jdent.2017.09.011. Epub 2017 Sep 27. PMID 28962842
- [Result] Panpisut P, Toneluck A. Monomer conversion, dimensional stability, biaxial flexural strength, and fluoride release of resin-based restorative material containing alkaline fillers. Dent Mater J. 2020 Aug 2;39(4):608-615. doi: 10.4012/dmj.2019-020. Epub 2020 Feb 7. PMID 32037385
- [Result] Swift EJ Jr, Perdigao J, Heymann HO, Wilder AD Jr, Bayne SC, May KN Jr, Sturdevant JR, Roberson TM. Eighteen-month clinical evaluation of a filled and unfilled dentin adhesive. J Dent. 2001 Jan;29(1):1-6. doi: 10.1016/s0300-5712(00)00050-6. PMID 11137632
- [Result] Vallittu PK, Boccaccini AR, Hupa L, Watts DC. Bioactive dental materials-Do they exist and what does bioactivity mean? Dent Mater. 2018 May;34(5):693-694. doi: 10.1016/j.dental.2018.03.001. Epub 2018 Mar 20. No abstract available. PMID 29571660
- [Derived] Mustafa K, Alfakhry G, Milly H. Periodontal Evaluation for a New Alkasite Restorative Material in Noncarious Cervical Lesions: A Randomized-Controlled Clinical Trial. Clin Exp Dent Res. 2024 Dec;10(6):e70025. doi: 10.1002/cre2.70025. PMID 39400529